CLINICAL TRIAL: NCT03277222
Title: HAND IN Insulin-001: Intranasal Treatment of HIV-associated Neurocognitive Disorders
Brief Title: Intranasal Treatment of HIV-associated Neurocognitive Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to find further eligible participants
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Alberta (Other); Epidemiology Coordinating and Research Centre, Canada (Other)
Responsible Party: Principal Investigator, John Gill, Medical Director, Southern Alberta Clinic, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB17-0104; Control# 204512 (Other: Health Canada)
Record Dates: First submitted 2017-08-28; First posted 2017-09-08 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: HIV Associated Neurocognitive Disorder (HAND)
Keywords: Neurocognitive impairment; HIV-1; Intranasal insulin; Neurocognitive Disorder; Cognition; Memory
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: Arm 1: Drug: IN insulin Dose: Twice daily IN insulin R at 40 IU (n=10) twice daily using a nasal delivery device. IN insulin R will be administered twice daily.
  Arm 2: Drug: Sterile Saline placebo Dose: Placebo (Sterile Saline placebo, matched volume; (n=10) twice daily using nasal delivery device.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a prospective dose-ranging double-blinded pilot study over 4 months. At enrolment, participants and their physicians will be blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IN insulin 40 IU (Active Comparator): Drug: IN insulin Dosage form: intranasal Dose: 40 IU Frequency: bid Duration: 16 weeks
  Interventions: Biological: IN insulin
- IN Sterile Saline (Placebo Comparator): Drug: Sterile Saline Dosage form: intranasal Frequency: bid Duration: 16 weeks
  Interventions: Biological: Sterile Saline placebo

INTERVENTIONS:
Biological: IN insulin — IN insulin twice daily taken after breakfast and again after dinner using the nasal delivery device.
  Other Names: Intranasal Humulin R
  Arms: IN insulin 40 IU
Biological: Sterile Saline placebo — Sterile Saline placebo twice daily taken after breakfast and again after dinner using the nasal delivery device.
  Arms: IN Sterile Saline

SUMMARY:
This study aims to see whether intranasal insulin is an effective treatment for problems with memory, concentration, slowed thinking, or any other cognitive function in people living with HIV/AIDS. This group of signs and symptoms are called 'HIV-associated neurocognitive disorders' or HAND. HAND can affect people living with HIV/AIDS even when they receive potent anti-HIV treatments. Treatment of HAND by specific medication or other means is not yet available. Intranasal insulin treatment has virtually no side-effects, and has already been tested in people with Alzheimer's disease, where it showed beneficial effects on memory, mood and quality of life

DETAILED DESCRIPTION:
This study is designed as a prospective, double-blinded pilot study of intranasal (IN) insulin versus placebo in people with HAND (n = 20) on stable ART medication. Participants will be randomly assigned to one of two groups: 40 IU IN insulin R twice daily, or matched-volume placebo, which will be administered twice daily, taken after breakfast and again after dinner using a nasal delivery device. Serum glucose will be tested for hypoglycemia one hour after the initial administration of IN insulin or placebo and after administration at Weeks 1, 2, and 3. If the dose is tolerated and no side effects are reported the participant will continue in the study. If the dose is not tolerated due to hypoglycemia then the participant will be withdrawn from the study.

The objectives of this study are as follows:

Primary: Determine if IN insulin treatment administered twice daily for 4 months reduces overall neurocognitive deficits (based on the global z-score in people with HAND).

Secondary: Measure effects of IN insulin on individual neuropsychological domains (e.g., memory, processing speed, executive functions, motor functions) and on HAND disease progression; Define impacts of IN insulin on quality of life and mood in people with HAND; Investigate IN insulin's effects on HAND biomarker profiles in urine and blood.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Maintained on stable ART for ≥6 months (defined as undetectable viral load)
* HAND-MND or -ANI diagnosis with evidence of clinical onset or progression within the prior 2 years, based on established criteria
* Currently followed at the Southern Alberta Clinic (SAC; Calgary, AB, Canada)

Exclusion Criteria:

* HAND with a) changed dose of any medication for HIV-1 infection with a corresponding increase in viral load (e.g., ART), or b) secondary therapies for HAND (e.g., memantine, amphetamines).
* Advanced liver, renal or lung disease, cancer or diabetes requiring insulin
* Secondary diagnosis of neurocognitive impairment or other major neuropsychiatric illness such as epilepsy, Alzheimer's or Parkinson's diseases, major depression (PHQ-9 score >10), or schizophrenia
* Central nervous system lesion (diagnosed by neuroimaging) that may impair cognition
* Previous allergic reaction to insulin or any of the carrier components.
* Education < 9 years or inability to read and write English fluently
* Uncontrolled HIV-1 or hepatitis C co-infection
* Inability to perform NP or questionnaire measures, functional illiteracy
* Past or current substance abuse that could interfere with the study assessments as determined by the PI
* Marijuana use on the day of NP testing
* Uncontrolled cardiovascular disease (hypertension, coronary or peripheral artery disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
Change in Global Neurocognitive Performance from Baseline | 18 weeks
  Change in overall neurocognitive function as measured by the global z score. The global z score is one measurement calculated as the average of z scores from each domain tested.

SECONDARY OUTCOMES:
Change from Baseline in Neurocognitive Performance: Memory | 18 weeks
  Change from baseline in the overall z score for the memory domain, calculated as the average of z scores from: Hopkins Verbal Learning Test, Logical Memory Test, and Brief Visual Memory Test (immediate and delayed recall).
Change from Baseline in Neurocognitive Performance: Executive Function | 18 weeks
  Change from baseline in the overall z score for the executive function domain, calculated as the average of z scores from: D-KEFS Trail-making Task (Letter-Switching) and Color-Word Interference (Stroop).
Change from Baseline in Neurocognitive Performance: Attention | 18 weeks
  Change from baseline in the overall z score for the attention domain, calculated as the average of z scores from: Symbol Digit Modalities Test, D-KEFS Trail-making Test (Number), and Color-Word Interference (Color and Word Reading).
Change from Baseline in Neurocognitive Performance: Motor Function | 18 weeks
  Change from baseline in the overall z score for the motor function domain, calculated as the average of z scores from: grooved pegboard completion times for dominant and non-dominant hands.
Change from Baseline in Neurocognitive Performance: Language | 18 weeks
  Change from baseline in the overall z score for the language domain, calculated as the average of z scores from: D-KEFS Letter and Category Verbal Fluency Tasks

OTHER OUTCOMES:
Change from baseline in HQoL questionnaire score | 18 weeks
  Change from baseline in health-related quality of life (HQoL) questionnaire score
Change from baseline in the PHQ-9 Questionnaire score | 18 weeks
  Change in the Patient Health Questionnaire-9 (PHQ-9) depressive symptoms score.
Change from Baseline in the Frailty Index Score - questionnaire and clinic assessment | 16 weeks
  Change in the overall Frailty Index score measured from baseline to Week 8.
Change from Baseline HAND inflammasome biomarker laboratory result profile | 16 weeks
  Change in inflammasome biomarker laboratory result profile between baseline and week 16.
Change from Baseline HAND metabolomics biomarker laboratory result profile | 16 weeks
  Change in metabolomics biomarker laboratory result profile between baseline and week 16.
Change from Baseline plasma HIV-1 viral load laboratory result | 16 weeks
  Change in plasma HIV-1 viral load between baseline and week 16.
Change from Baseline blood CD4 T-cell count laboratory result | 16 weeks
  Change in blood CD4 T-cell count between baseline and week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Power, MD, FRCPC, Principal Investigator — University of Alberta; Michael J Gill, MBChB FACP, Principal Investigator — University of Calgary
Locations (1):
- Southern Alberta Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antinori A, Arendt G, Becker JT, Brew BJ, Byrd DA, Cherner M, Clifford DB, Cinque P, Epstein LG, Goodkin K, Gisslen M, Grant I, Heaton RK, Joseph J, Marder K, Marra CM, McArthur JC, Nunn M, Price RW, Pulliam L, Robertson KR, Sacktor N, Valcour V, Wojna VE. Updated research nosology for HIV-associated neurocognitive disorders. Neurology. 2007 Oct 30;69(18):1789-99. doi: 10.1212/01.WNL.0000287431.88658.8b. Epub 2007 Oct 3. PMID 17914061
- [Background] Pandya R, Krentz HB, Gill MJ, Power C. HIV-related neurological syndromes reduce health-related quality of life. Can J Neurol Sci. 2005 May;32(2):201-4. doi: 10.1017/s0317167100003978. PMID 16018155
- [Background] Yeung H, Krentz HB, Gill MJ, Power C. Neuropsychiatric disorders in HIV infection: impact of diagnosis on economic costs of care. AIDS. 2006 Oct 24;20(16):2005-9. doi: 10.1097/01.aids.0000247565.80633.d2. PMID 17053346
- [Background] Vivithanaporn P, Heo G, Gamble J, Krentz HB, Hoke A, Gill MJ, Power C. Neurologic disease burden in treated HIV/AIDS predicts survival: a population-based study. Neurology. 2010 Sep 28;75(13):1150-8. doi: 10.1212/WNL.0b013e3181f4d5bb. Epub 2010 Aug 25. PMID 20739646
- [Background] Mamik MK, Asahchop EL, Chan WF, Zhu Y, Branton WG, McKenzie BA, Cohen EA, Power C. Insulin Treatment Prevents Neuroinflammation and Neuronal Injury with Restored Neurobehavioral Function in Models of HIV/AIDS Neurodegeneration. J Neurosci. 2016 Oct 12;36(41):10683-10695. doi: 10.1523/JNEUROSCI.1287-16.2016. PMID 27733618
- [Background] Boisse L, Gill MJ, Power C. HIV infection of the central nervous system: clinical features and neuropathogenesis. Neurol Clin. 2008 Aug;26(3):799-819, x. doi: 10.1016/j.ncl.2008.04.002. PMID 18657727
- [Background] Fujiwara, E., Gill, J.M. & Power, C. Risk Factors for HIV-Associated Neurocognitive Disorders (HAND) in a Canadian Cohort (P1.321). Neurology 86 P1.321 (2016).
- [Background] McCombe JA, Vivithanaporn P, Gill MJ, Power C. Predictors of symptomatic HIV-associated neurocognitive disorders in universal health care. HIV Med. 2013 Feb;14(2):99-107. doi: 10.1111/j.1468-1293.2012.01043.x. Epub 2012 Sep 20. PMID 22994556
- [Background] Grant I, Franklin DR Jr, Deutsch R, Woods SP, Vaida F, Ellis RJ, Letendre SL, Marcotte TD, Atkinson JH, Collier AC, Marra CM, Clifford DB, Gelman BB, McArthur JC, Morgello S, Simpson DM, McCutchan JA, Abramson I, Gamst A, Fennema-Notestine C, Smith DM, Heaton RK; CHARTER Group. Asymptomatic HIV-associated neurocognitive impairment increases risk for symptomatic decline. Neurology. 2014 Jun 10;82(23):2055-62. doi: 10.1212/WNL.0000000000000492. Epub 2014 May 9. PMID 24814848
- [Background] Sacktor N, Skolasky RL, Seaberg E, Munro C, Becker JT, Martin E, Ragin A, Levine A, Miller E. Prevalence of HIV-associated neurocognitive disorders in the Multicenter AIDS Cohort Study. Neurology. 2016 Jan 26;86(4):334-40. doi: 10.1212/WNL.0000000000002277. Epub 2015 Dec 30. PMID 26718568
- [Background] Nightingale S, Winston A, Letendre S, Michael BD, McArthur JC, Khoo S, Solomon T. Controversies in HIV-associated neurocognitive disorders. Lancet Neurol. 2014 Nov;13(11):1139-1151. doi: 10.1016/S1474-4422(14)70137-1. PMID 25316020
- [Background] Letendre S, Marquie-Beck J, Capparelli E, Best B, Clifford D, Collier AC, Gelman BB, McArthur JC, McCutchan JA, Morgello S, Simpson D, Grant I, Ellis RJ; CHARTER Group. Validation of the CNS Penetration-Effectiveness rank for quantifying antiretroviral penetration into the central nervous system. Arch Neurol. 2008 Jan;65(1):65-70. doi: 10.1001/archneurol.2007.31. PMID 18195140
- [Background] Hyun E, Ramachandran R, Hollenberg MD, Vergnolle N. Mechanisms behind the anti-inflammatory actions of insulin. Crit Rev Immunol. 2011;31(4):307-40. doi: 10.1615/critrevimmunol.v31.i4.30. PMID 21899513
- [Background] Benedict C, Hallschmid M, Hatke A, Schultes B, Fehm HL, Born J, Kern W. Intranasal insulin improves memory in humans. Psychoneuroendocrinology. 2004 Nov;29(10):1326-34. doi: 10.1016/j.psyneuen.2004.04.003. PMID 15288712
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Rosenbloom MH, Barclay TR, Pyle M, Owens BL, Cagan AB, Anderson CP, Frey WH 2nd, Hanson LR. A single-dose pilot trial of intranasal rapid-acting insulin in apolipoprotein E4 carriers with mild-moderate Alzheimer's disease. CNS Drugs. 2014 Dec;28(12):1185-9. doi: 10.1007/s40263-014-0214-y. PMID 25373630
- [Background] Claxton A, Baker LD, Wilkinson CW, Trittschuh EH, Chapman D, Watson GS, Cholerton B, Plymate SR, Arbuckle M, Craft S. Sex and ApoE genotype differences in treatment response to two doses of intranasal insulin in adults with mild cognitive impairment or Alzheimer's disease. J Alzheimers Dis. 2013;35(4):789-97. doi: 10.3233/JAD-122308. PMID 23507773
- [Background] Claxton A, Baker LD, Hanson A, Trittschuh EH, Cholerton B, Morgan A, Callaghan M, Arbuckle M, Behl C, Craft S. Long-acting intranasal insulin detemir improves cognition for adults with mild cognitive impairment or early-stage Alzheimer's disease dementia. J Alzheimers Dis. 2015;44(3):897-906. doi: 10.3233/JAD-141791. PMID 25374101
- [Background] Reger MA, Watson GS, Green PS, Wilkinson CW, Baker LD, Cholerton B, Fishel MA, Plymate SR, Breitner JC, DeGroodt W, Mehta P, Craft S. Intranasal insulin improves cognition and modulates beta-amyloid in early AD. Neurology. 2008 Feb 5;70(6):440-8. doi: 10.1212/01.WNL.0000265401.62434.36. Epub 2007 Oct 17. PMID 17942819
- [Background] Shemesh E, Rudich A, Harman-Boehm I, Cukierman-Yaffe T. Effect of intranasal insulin on cognitive function: a systematic review. J Clin Endocrinol Metab. 2012 Feb;97(2):366-76. doi: 10.1210/jc.2011-1802. Epub 2011 Dec 7. PMID 22162476
- [Background] Asahchop EL, Akinwumi SM, Branton WG, Fujiwara E, Gill MJ, Power C. Plasma microRNA profiling predicts HIV-associated neurocognitive disorder. AIDS. 2016 Aug 24;30(13):2021-31. doi: 10.1097/QAD.0000000000001160. PMID 27191977
- [Background] Lenart N, Brough D, Denes A. Inflammasomes link vascular disease with neuroinflammation and brain disorders. J Cereb Blood Flow Metab. 2016 Oct;36(10):1668-1685. doi: 10.1177/0271678X16662043. Epub 2016 Aug 2. PMID 27486046
- [Background] Walsh JG, Muruve DA, Power C. Inflammasomes in the CNS. Nat Rev Neurosci. 2014 Feb;15(2):84-97. doi: 10.1038/nrn3638. Epub 2014 Jan 8. PMID 24399084
- [Background] Kim DH, Jewison DL, Milner GR, Rourke SB, Gill MJ, Power C. Neurocognitive symptoms and impairment in an HIV community clinic. Can J Neurol Sci. 2001 Aug;28(3):228-31. doi: 10.1017/s0317167100001372. PMID 11513341
- [Background] Koenig N, Fujiwara E, Gill MJ, Power C. Montreal Cognitive Assessment Performance in HIV/AIDS: Impact of Systemic Factors. Can J Neurol Sci. 2016 Jan;43(1):157-62. doi: 10.1017/cjn.2015.306. Epub 2015 Dec 4. PMID 26635008
- [Background] Fujiwara E, Tomlinson SE, Purdon SE, Gill MJ, Power C. Decision making under explicit risk is impaired in individuals with human immunodeficiency virus (HIV). J Clin Exp Neuropsychol. 2015;37(7):733-50. doi: 10.1080/13803395.2015.1057481. Epub 2015 Jul 24. PMID 26207583
- [Background] Justice AC, McGinnis KA, Atkinson JH, Heaton RK, Young C, Sadek J, Madenwald T, Becker JT, Conigliaro J, Brown ST, Rimland D, Crystal S, Simberkoff M; Veterans Aging Cohort 5-Site Study Project Team. Psychiatric and neurocognitive disorders among HIV-positive and negative veterans in care: Veterans Aging Cohort Five-Site Study. AIDS. 2004 Jan 1;18 Suppl 1:S49-59. PMID 15075498
- [Background] Crane HM, Van Rompaey SE, Dillingham PW, Herman E, Diehr P, Kitahata MM. A single-item measure of health-related quality-of-life for HIV-infected patients in routine clinical care. AIDS Patient Care STDS. 2006 Mar;20(3):161-74. doi: 10.1089/apc.2006.20.161. PMID 16548713
- [Background] Power C, Gill MJ, Johnson RT. Progress in clinical neurosciences: The neuropathogenesis of HIV infection: host-virus interaction and the impact of therapy. Can J Neurol Sci. 2002 Feb;29(1):19-32. doi: 10.1017/s0317167100001682. PMID 11858531
- [Background] Van Marle G, Rourke SB, Zhang K, Silva C, Ethier J, Gill MJ, Power C. HIV dementia patients exhibit reduced viral neutralization and increased envelope sequence diversity in blood and brain. AIDS. 2002 Sep 27;16(14):1905-14. doi: 10.1097/00002030-200209270-00007. PMID 12351950
- [Background] Skinner S, Adewale AJ, DeBlock L, Gill MJ, Power C. Neurocognitive screening tools in HIV/AIDS: comparative performance among patients exposed to antiretroviral therapy. HIV Med. 2009 Apr;10(4):246-52. doi: 10.1111/j.1468-1293.2008.00679.x. Epub 2009 Jan 23. PMID 19187172
- [Background] McCombe JA, Auer RN, Maingat FG, Houston S, Gill MJ, Power C. Neurologic immune reconstitution inflammatory syndrome in HIV/AIDS: outcome and epidemiology. Neurology. 2009 Mar 3;72(9):835-41. doi: 10.1212/01.wnl.0000343854.80344.69. PMID 19255411
- [Background] Sacktor, N., et al. Paroxetine and Fluconazole Therapy for HAND: A Double-Blind, Placebo-Controlled Trial. Conference on retroviruses and opportunistic infections. 2016 Boston MA USA Sesssion O-12 Abstract 146(2016).
- [Background] Power C, Boisse L, Rourke S, Gill MJ. NeuroAIDS: an evolving epidemic. Can J Neurol Sci. 2009 May;36(3):285-95. doi: 10.1017/s0317167100007009. PMID 19534327